CLINICAL TRIAL: NCT04512092
Title: Affiliative Mentality in Residential Youth Care: A Cluster Randomized Trial of a Compassionate Mind Training Program With Caregivers
Brief Title: The Efficacy of a Compassionate Mind Training Program With Caregivers of Residential Youth Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Laura Filipa Seiça Matias Santos, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/132327/2017; SFRH/BD/132327/2017 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2020-08-06; First posted 2020-08-13 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Compassion
Keywords: Residential Care; Compassionate Mind Training; Caregivers; Children and adolescents at risk; Compassion
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMT-C group (Experimental): Compassion Mind Training for Caregivers (CMT-C) is a 12-session structured program to be delivered in a group format, aiming to cultivate a compassionate-self and compassionate care practices in residential youth care.
  Interventions: Behavioral: Compassionate Mind Training for Caregivers
- Control group (No Intervention): This group did not receive any mind training or group intervention during the study.

INTERVENTIONS:
Behavioral: Compassionate Mind Training for Caregivers — CMT-C is a 12-session group program, each lasting about 2,5 hours, which run on a weekly basis. The program is organized across 3 modules: 1) Our mind according to a compassion-based approach (to provide insight into the evolved and socially shaped mind and the affect regulation systems); 2) Compassionate mind training (understanding and cultivating the attributes and competencies of compassion in its three flows, and addressing its fears); and 3) final session (revising key information and practices and its application to the RCH practices/routines). Its sessions have the following structure: 1) Check-in (grounding exercise, reviewing the previous session, sharing the weekly practice); 2) Exploration of the session theme (psychoeducation and experiential practices followed by group opportunities for share experiences and discussion); 3) Check-out (session summary and application to the self, youths and RCH practices, weekly practice challenge, session evaluation, session take-off).
  Arms: CMT-C group

SUMMARY:
This clinical trial aims to improve the quality of the care provided in residential youth care, through a Compassionate Mind Training (CMT-C) program targeted to caregivers. The promotion of an affiliative mentality of caring, warmth and affection in the residential care setting is operationalized through the development of a compassionate-self and compassionate care skills. A cluster randomized trial with a control group was carried out in order to test the efficacy of a 12-session Compassionate Mind Training Program to caregivers of residential youth care in increasing compassion, self-compassion, social safeness, emotional climate, empathy, emotion regulation, satisfaction with life, and resiliency and in reducing self-criticism, fears of compassion as well as stress, burnout, anxiety and depression. Youths in residential care were also assessed as informants, thought self-reported questionnaires on current experiences of warmth and safeness, social safeness, emotional climate, positive and negative affect. The organizational impact was assessed via focus groups. It is hypothesized that the CMT-C would produce significant improvements in outcome measures, when comparing caregivers who receive the CMT-C with those in the control group. It is expected that after the training, caregivers will present a greater sensibility to their own and others suffering and motivation to relieve it, exhibiting and experiencing empathic responses. Consequently, it is also expected that youths in care perceive more warmth and safeness experiences with caregivers and a more secure and safe emotional climate in the residential care home.

DETAILED DESCRIPTION:
This was a Cluster Randomized Trial with a control group carried out in twelve Portuguese Residential Youth Care facilities. It aimed to test the efficacy of a group-based Compassionate Mind Training program (CMT-C) targeted to caregivers, in promoting significant changes both in caregivers and adolescents in residential youth care. This trial was carried out in accordance with the ethical principles of the Declaration of Helsinki and the applicable national laws and regulations. The ethics committee of the Faculty of Psychology and Educational Sciences of the University of Coimbra approved the study's procedures.

Since CMT-C is targeted for residential care homes' (RCH) teams, for practical reasons (to maximize time and human resources) and to avoid contamination, the unit of randomization was the RCH (i.e., cluster), hence a cluster randomized design was followed according CONSORT guidelines. From the 32 RCH within the Centre region of Portugal, 19 RCH obeying to cluster eligibility criteria were invited to participate. Twelve RCH agreed to enter the trial. Their caregivers and adolescents, who were eligible for the study, were informed of the goals and procedures of this research, and invited to voluntarily participate. No incentives were offered for participation. Written informed consent were sought at the cluster level (from the board of each RCH), and at the individual level to caregivers and adolescents (and their legal guardians), before the randomization occurred. Adolescents aged between 14 and 16 YO, gave informed assent, while the older than 16 YO will give written informed consent. A written informed consent was also gathered from guardians/legal representatives of all adolescent participants under 18 YO. The anonymity of all participants responses was guaranteed, with the use of respondent-specific codes, which were also used to link the data from one time point to the other. Data was collectively collected in each RCH with the presence of an independent researcher, in order to answer any questions and ensure confidentiality. All participants (caregivers and adolescents) were assessed through self-report measures 5 times across 12 months. Specifically, participants were assessed 3 months before the beginning of the CMT-C (Baseline 0 - time 0), before the first session of the program (baseline 1 - time 1), right after its terminus (i.e., post-treatment assessment - time 2), and 3 and 6 months after intervention terminus (follow-up 1 and 2 - time 3 and time 4). Participants in the control group were assessed with the same time intervals as those in intervention group.

After the first baseline assessment, a computer-generated randomization was conducted at the cluster level, following a completely randomized design. Each RCH (i.e., cluster) was randomly assigned to one of two conditions: CMT-C and control group. Six RCH were allocated in the experimental group and received the TMC for caregivers, the remaining 6 constituted the control group. Caregivers in the treatment group attended the CMT-C for about 12 weeks. The CMT-C consisted of twelve, 2.5-hr weekly group sessions, delivered in each RCH to a group of 7 to 10 participants. Caregivers in the control group did not received any mind training or group intervention.

After post-treatment assessments, focus groups were carried out with the caregivers allocated in the CMT-C group, in order to enrich understanding about the participants' experience with the intervention and their perception of change at 3 different levels (individual, interindividual and organizational).

Treatment integrity were ensured through: a) specific treatment manuals; b) direct training of the therapist; c) supervision; and d) assessment of adherence and competence through an integrity rating scale.

Treatment effects will be analyzed following an intention-to-treat analysis using Latent Growth Curve Models (LGCM). The intercept (i.e., initial status) and slope (i.e., change over time) will be modeled as latent variables from longitudinal data (T0 to T4). Per-protocol analysis will also be carried out to investigate treatment effects in completers. Moderator (e.g., clusters) effects will also be tested with Conditional LGCM, and will be included as predictors of change over time in the outcome measures. Nested qualitative evaluation with thematic analysis will be carried out after the last follow-up.

ELIGIBILITY:
Eligibility criteria for clusters:

Inclusion criteria: Residential care homes (RCH) in the Centre region of Portugal, receiving adolescents (both genders) aged between 12 and 25 YO.

Exclusion criteria: RCH mostly receiving children or specialized in mental and behavioural disorders/substance abuse problems will be excluded (to control for mental health treatments delivered in these RCH).

Eligibility criteria for participants:

Inclusion criteria for caregivers: Professionals working in RCH and directly interacting with the adolescents on a regular basis.

Inclusion criteria for adolescents: have entered in the RCH at least 1-month before the study's onset (adjustment time); aged between 12 and 25 YO.

Exclusion criteria for adolescents: cognitive impairment; remaining in residential care for less than 9 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Change of Compassion | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Compassion Scale (CS; Pommier, 2011; Portuguese version by Sousa, Castilho, Vieira, Vagos, & Rijo, 2017). The CS is a 24-item self-report scale that measures compassion for others. Participants answered each item according to how frequently they feel and act towards others, using a 5-point Likert scale (1 = almost never, to 5 = almost always). In the Portuguese version, a CFA revealed the existence of six subscales and two higher-order factors: Compassion (comprising the positive subscales: Kindness, Common Humanity, Mindfulness) and Disconnectedness (comprising the negative subscales: Indifference, Separation and Disengagement), which represent a positive and a negative valence of compassion.
Change of Self-Compassion | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Self-Compassion Scale (SCS; Neff, 2003; Portuguese version by Castilho, Pinto-Gouveia & Duarte, 2015). The SCS is a 26 self-reported scale which addresses self-compassion and instructs participants to answer its items, rated in a 5-point Likert scale (1 = almost never, to 5 = almost always), regarding "how I typically act towards myself in difficult times". In the original version, the scale has a total score and six subscales (Self-Kindness; Self-Judgement; Common Humanity; Isolation; Mindfulness; and Over-Identification). The Portuguese version tested a two-factor model, finding that a Self-Compassionate attitude (comprising the positive subscales: Self-Kindness, Common Humanity, Mindfulness) and Self-Critical attitude (comprising the negative subscales: Self-Judgement, Isolation and Over-Identification).
Change of Fears of Compassion | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Fears of Compassion Scales (FCS; Gilbert, McEwan, Matos, & Rivis, 2011; Portuguese version by Matos, Pinto-Gouveia, Duarte, & Simões, 2011). The FCS integrates three self-reported scales designed to assess fears of being compassionate toward others (10 items), receiving compassion from others (13 items) and being self-compassionate (15 items). The items were rated on a 5-point Likert scale (0 = Do not agree at all, to 4 = Completely agree).
Change of Social Safeness | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Social Safeness and Pleasure Scale (SSPS; Gilbert et al., 2009; Portuguese version by Dinis, Castilho, Xavier, & Pinto-Gouveia, 2008). The SSPS is an 11-item unidimensional self-reported scale that assesses the frequency with which individuals experience positive feelings in their social relationships, as well as, they experience the world as a safe and soothing place. Items are rated through a 5-point Likert scale (1 =almost never, to 5=almost always).
Change of Emotional Climate at the workplace | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Emotional Climate in Organizations Scale Adults (ECOS-A; Albuquerque et al., 2018). The ECOS-A is a 30-item self-report scale, aiming to assess how workers felt and behaved at their workplace, over the past two weeks. This scale has two parts (i.e., emotions and motives) with 15 items each. Each one is divided into 3 subscales, with 5 items, referring to the three affect's regulation systems: the threat system, the soothing system and the drive system. All items are answered according to a 5-points Likert's scale (0 =Never, to 4= Always).

SECONDARY OUTCOMES:
Emotion regulation | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski, Kraaij, & Spinhoven, 2002; Portuguese version by Castro et al., 2013). CERQ is a 36 items self-report questionnaire designed to measure specific cognitive emotion regulation used in response to the experience of threatening or stressful events. It has nine subscales, each one corresponding to one cognitive emotion regulation strategy: Self-Blame (SB), Rumination (R), Positive Refocusing (PRF), Planning (P), Other-Blame (OB), Catastrophizing (C), Putting into Perspective (PIP), Positive Reappraisal (PRP) and Acceptance (A). Each subscale has 4 items, answered on a five-point Likert scale ranging from 1 (almost never) to 5 (almost always).
Mental Health Symptoms | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Depression, Anxiety and Stress Scale (DASS-21; Lovibond & Lovibond, 1995; Portuguese version by Pais-Ribeiro, Honrado & Leal, 2004). DASS-21 is a 21 items self-report measure designed to assess three dimensions of psychopathological symptoms: depression, anxiety, and stress. Items are rated using a four-point Likert scale for frequency (ranging from 0=Does not apply to me at all to 3 =Applied to me very much or most of the time).
Professional Quality of Life | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Professional Quality of Life Scale, version 5 (ProQOL-5; Stamm, 2010; Portuguese version by Carvalho, 2011). The ProQOL is a 30-item self-report measure composed by three subscales: compassion satisfaction (CS), burnout (BO) and secondary traumatic stress (STS). Participants are instructed to indicate how frequently each item was experienced in the previous 30 days, on a 5-point Likert scale (from 1 = never to 5 = very often).
Empathy | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Interpersonal Reactivity Index (IRI; Davis, 1983; Portuguese version by Limpo, Alves & Castro, 2010). IRI is a 24-item self-reported scale, aiming to measure perspective taking, empathic concern and fantasy. Perspective taking is considered a cognitive component of empathy, while empathic concern and personal distress are considered the affective component. Respondents are instructed to rate how well each statement describes them on a 5- point Likert scale (from 0 = not well to 4 = very well).
Resilience | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Resilience Scale (RS; Wagnild & Young, 1993; Portuguese version by Pinheiro & Matos, 2013). RS is a 14-item self-reported scale aiming to assess resiliency. Respondents are instructed to rate how well each statement describes them on a 7- point Likert scale (from 1 = Completely disagree, to 7 = Completely agree).
Satisfaction with life | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers reported on the Satisfaction With Life Scale (SWLS; Diener, Emmons, Larsen, & Griffin, 1985; Portuguese version by Simões, 1992) SWLS is a 5-item scale that measures the cognitive-judgmental aspects of general life satisfaction. Each item is scored from 1 to 7 on a Likert-type scale ranging from strongly disagree to strongly agree.
Positive and negative affect | baseline; 3 months; 6 months; 9 months; 12 months
  Caregivers and adolescents reported on the Positive and Negative Affect Schedule (PANAS; Watson et al., 1988; Portuguese version for adolescents by Galinha & Pais-Ribeiro, 2005). PANAS is a 20-item self-report scale designed to assess two mood states: positive affect and negative affect. Each subscale is composed by 10 items, that describe feelings and emotions. Participants are asked to rate the severity and frequency of these feelings and emotions in the last few weeks, using a 5-point Likert scale (1=nothing or very slightly, to 5=extremely).
Warmth and Safeness experiences | baseline; 3 months; 6 months; 9 months; 12 months
  Adolescents reported on the Current Experiences of warmth and safeness (CEWSS-A) (Santos, Sousa, Pinheiro & Rijo, 2020). The CEWSS-A is a 12-items self-report measure designed to assess the frequency in which adolescents feel emotional experiences of warmth, care, safeness with others, in the time period of the last two weeks. Items are answered using a Likert-scale response ranging from 0 (No, never) to 4 (Yes, most of the time).
Social safeness | baseline; 3 months; 6 months; 9 months; 12 months
  Adolescents reported on the Social Safeness and Pleasure Scale for Adolescents (SSPS-A; Gilbert et al., 2009; Portuguese version for adolescents by Castilho et al., 2015). The SSPS-A is an 11-item unidimensional self-reported scale that assesses the frequency with which individuals experience positive feelings in their social relationships, as well as, they experience the world as a safe and soothing place. Items are rated through a 5-point Likert scale (1 =almost never, to 5=almost always).
Emotional Climate in Residential Care Home | baseline; 3 months; 6 months; 9 months; 12 months
  Adolescents reported on the Emotional Climate in the Classroom Scale (ECCS; Albuquerque, Matos, Cunha, Galhardo, Palmeira, & Lima, 2018). ECCS is a 15-item self-report scale aiming to assess how adolescents feel in classroom over the past two weeks. This scale is divided into 3 subscales, which one with 5 items, describing different feelings associated to the three affect's regulation systems: the threat system, the soothing system and the drive system. Items are answered according to a Likert's scale, ranging from 0 "Never" to 4 "Always".
Internalizing and externalizing problems | baseline; 3 months; 6 months; 9 months; 12 months
  Adolescents reported on the Strengths and Difficulties Questionnaire (SDQ; Goodman, Meltzer, & Bailey, 1998; Portuguese version by Fleitlich et al., 2005). The self-report SDQ version has 25-items rated using a Likert-type response scale ranging from 0 (not true) to 2 (certainly true). It can be completed by young people aged 11-17 years and is organized into five subscales - emotional symptoms, conduct problems, hyperactivity/inattention difficulties, peer relationship problems and prosocial behaviors. SDQ bi-factor model - internalizing and externalizing has been extensively used.

OTHER OUTCOMES:
Focus groups for the assessement of organizational change | Two weeks after post-intervention assessments
  In order to enrich understanding about the participants' experience with the intervention and their perception of change, focus groups (FG) will be conducted 2 weeks after the final CMT-C session with the caregivers, who attended the CMT-C. The FG will be moderated by the researcher and an assistant, following a FG guide (Santos, Pinheiro & Rijo, 2019), composed by 12 open ended questions, regarding their experiences with CMT-C, learnings transfer, perception of change, impact and learning sustainability in residential care. The FG will be audio recorded and transcribed verbatim.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rijo, PhD, Study Director — CINEICC
Locations (1):
- Faculty of Psychology and Educational Sciencies, University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Santos L, Pinheiro MDR, Rijo D. The Effects of the Compassionate Mind Training for Caregivers on Professional Quality of Life and Mental Health: Outcomes from a Cluster Randomized Trial in Residential Youth Care Settings. Child Youth Care Forum. 2023 May 3:1-21. doi: 10.1007/s10566-023-09749-6. Online ahead of print. PMID 37360762